CLINICAL TRIAL: NCT01270048
Title: The Effect of Bunsimgi-eum(Fenxinqiyin) on the Chest Discomfort of Hwa-byung's Major Symptom : Randomized, Double-blinded, Placebo-control Trial
Brief Title: The Effect of Bunsimgieum on the Chest Discomfort of Hwa-byung's Major Symptom
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Sun-Tae. Kim, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B070057
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2009-09

CONDITIONS: Hwa-byung (Disorder)
Keywords: Hwa-byung, Bunsimgi-eum(Fenxinqiyin)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bunsimgieum extract (Experimental): * name of product: 'mild-x-gwarip'
  * standard code for item: 200005689
  * shape, type: extract(brown)
  * usage, content: adults;three times a day, each taken before or between meals
  * dose, standard: 2.5g for each sack, capsulated
  * storage : airtight container, stored in room temperature
  * expiration date : 36months after manufacture
  * macufacturing company: KyungBangnShinYak inc.
  Interventions: Drug: mild-ex-gwarip
- Placebo; corn flour, (Placebo Comparator): * raw material: total contents(500㎎); cornstarch 50.0%(250.0㎎), 당수화물 49.45%(247.25㎎), caramel pigment 0.5%(2.5㎎), SsangHwa fragrance 0.05%(0.25㎎)
  * shape, type: extract(brown)
  * usage, dose: adults: three times a day, 1 sack before or between meals
  * dose, standard: 2.5g for each sack, capsulated
  * storage : airtight container, stored in room temperature
  * expiration date : 36 months after manufacture
  * manufacturing company: KyungBangnShinYak inc.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: mild-ex-gwarip — three times a day, AC 30 min., 4 capsules taken each time (4capsules=2.5g), 8 weeks.
  Other Names: standard code for item: 200005689
  Arms: Bunsimgieum extract
Other: Placebo — three times a day, AC 30 min., 4 capsules taken each time (4capsules=2.5g), 8 weeks.
  Arms: Placebo; corn flour,

SUMMARY:
The purpose of this research is to examine the effect of Bunsimgi-eum on the chest discomfort of Hwa-byung's major symptom and develope and establish pattern identification system in Hwa-byung.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 20-65
* subjects who meet structured interview criteria for Hwa-Byung Diagnosis

Exclusion Criteria:

* duration of illness less than 6 months
* current or past history of delusions, hallucination
* past history of at least one manic episode, hypomanic episode, or mixed episode
* current or past history of alcohol abuse or alcohol dependence history
* taking substances(e.g. steroids) which might affect symptoms
* medical conditions(e.g. hyperthyroidism, hypothyroidism, heart disease) that might affect symptoms
* current with hepatoma, hepatic cirrhosis, chronic renal failure, congestive heart failure
* pregnancy, lactation, women not using medically accepted means of birth control
* considered not apt to carry out clinical trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In-Chul Jung, Ph.D, Principal Investigator — Oriental Hospital of Daejon University
Locations (1):
- Oriental Hospital of Daejon University, Daejeon, Choong-Chung-Do, South Korea